CLINICAL TRIAL: NCT04628429
Title: Autonomic Functions in Migraine Patients as a Function of Migraine Status and CGRP Inhibition
Brief Title: CGRP Inhibition, Autonomic Function, and Migraine
Acronym: CGRP-1
Status: Recruiting | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Prof. Christian Wöber, MD, Associate Professor, Medical University of Vienna
Other Study IDs: EK Nr:1910/2020
Record Dates: First submitted 2020-11-05; First posted 2020-11-13 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Episodic Migraine; Chronic Migraine
Keywords: Calcitonin gene-related peptide inhibition; Monoclonal antibodies; Autonomic function; Composite Autonomic Symptom Scale 31; Migraine Disability Assessment Scale; Depression Anxiety Stress Scales; Cardiovascular Autonomic Dysfunction; Headache Impact Questionnaire
MeSH Terms: interventions — erenumab; galcanezumab; fremanezumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Episodic Migraine: All patients who have been diagnosed with migraine without aura or migraine with aura according to the diagnostic criteria of the International Classification of Headache Disorders, third edition (ICHD-3) and have been unsuccessfully treated with first-line prophylactic medication
  Interventions: Drug: Erenumab; Drug: Galcanezumab; Drug: Fremanezumab
- Chronic Migraine: All patients who have been diagnosed with chronic migraine (≥15 headache days per month 8 of which with migrainous features) according to the diagnostic criteria of the International Classification of Headache Disorders, third edition (ICHD-3) and have been unsuccessfully treated with first-line prophylactic medication
  Interventions: Drug: Erenumab; Drug: Galcanezumab; Drug: Fremanezumab
- Healthy Control: Controls must be healthy (free of any diagnosed chronic disease, acute infection requiring medication, family history or personal history of migraine), chosen to be as similar as possible to migraine patients, in terms of age and sex.

INTERVENTIONS:
Drug: Erenumab — anti-CGRP-receptor monoclonal anti-body
  Other Names: Aimovig®
  Groups: Chronic Migraine; Episodic Migraine
Drug: Galcanezumab — anti-CGRP-ligand monoclonal anti-body
  Other Names: Emgality®
  Groups: Chronic Migraine; Episodic Migraine
Drug: Fremanezumab — anti-CGRP-ligand monoclonal anti-body
  Other Names: Ajovy®
  Groups: Chronic Migraine; Episodic Migraine

SUMMARY:
The purpose of this clinical study is to better understand the function of the autonomic nervous system in patients with migraine. We aim to understand whether the autonomic functions change depending on the migraine status (i.e. whether they are between or during attacks) and whether the CGRP monoclonal antibody (mAb) class of drugs affects the autonomic functions. The aim is not to investigate the effect of CGRP-mAb on migraine frequency. Calcitonin gene-related peptide (CGRP) is a neurotransmitter in the nervous system that plays an essential role in the development of migraine headache. Monoclonal antibodies can block the function of this messenger substance. Several studies have shown that this blockade leads to a reduction in the frequency of migraine.

In addition to its role in migraine, CGRP also acts on the blood vessels and the autonomic nervous system. The autonomic nervous system is responsible for everything we have no control over in our body. This includes everything from heart rate and blood pressure to our digestion.

DETAILED DESCRIPTION:
Background:

Headache disorders are among the leading illnesses contributing to the Global Burden of Disease. They are so common, that they rank second in prevalence and years lived with disability. Additionally, headache disorders are the second-ranked cause of years lived with disability in females, worldwide. Migraines are so prevalent in human history that there exist records from the ancient Egyptians documenting symptoms of attacks.

Migraines are classified by the International Headache Society in their International Classification of Headache Disorders 3 (ICHD-3) guidelines as: migraine without aura, migraine with aura, chronic migraine, and probable migraine. They are considered episodic if headache is present on fewer than 15 days per month; or chronic if headache occurs "on 15 or more days/month for more than 3 months, which, on at least 8 days/month, has the features of migraine headache". Until now, researchers have made numerous connections between migraines and the autonomic symptoms that manifest both ictally and interictally. Research, using standardized autonomic tests, has improved our ability to evaluate these symptoms. Furthermore, strides have been made to map migraine attacks and visualize them. Finally, research directed towards the molecular mechanism of these attacks has also yielded results.

Current recommendations for pharmacological migraine treatment comprise abortive drugs (i.e. non-opioid analgesics and triptans) and prophylactic medication (e.g. beta-blockers, calcium-channel blockers, antidepressants, anti-seizure medications and onabotulinumtoxin A). None of these prophylactic drugs were specifically developed against migraine. Their dosages must be slowly increased, since these medications can lead to fatigue, depression, nausea, insomnia, decreased libido, along with many other side effects specific to the individual modalities. Therefore, a more favorable treatment is required.

Molecular evidence is accumulating that calcitonin gene-related peptide (CGRP) contributes greatly to this pathophysiology. In tandem, evidence of CGRP's role in other physiological mechanisms has also been elucidated. These include roles in: vasodilation, cardioprotection, blood pressure regulation, sepsis, wound healing, bone re-growth, among others. The majority of CGRP is sequestered at the trigeminal level; however, it is released from both peripheral and central nerve terminals. As such, investigation of parasympathetic - and reciprocally, the sympathetic - autonomic nervous system (ANS) pathways are of particular interest. It is, however, CGRP's connection to migraines which has, consequently, led to the development of several CGRP receptor antagonists, an anti-CGRP-receptor monoclonal anti-body (mAb) and several anti-CGRP-ligand mAbs.

Only recently have anti-CGRP antibodies been approved by the European Medicines Agency. There are three prophylactic pharmaceutical options targeting CGRP currently available and reimbursed in Austria. Erenumab (Aimovig® - anti-receptor) is available since September 2018, Galcanezumab (Emgality® - anti-ligand) since March 2019 and Fremanezumab (Ajovy® - anti-ligand) since May 2019. Randomized controlled trials are also ongoing for Eptinezumab (anti-ligand). The largest benefit provided by anti-CGRP monoclonal antibodies is that they are relatively well-tolerated - shown to reduce the frequency of attacks experienced by the patient each month. As such, CGRP-related monoclonal antibodies are being increasingly utilized; however, there is a very limited amount of exogenous medication that does not have unwanted interactions once administered into the body.

In randomized, placebo-controlled studies on the efficacy and tolerability of anti-CGRP monoclonal antibodies (ant-CGRP-mAbs), no serious side effects were found. Those that were found and are provided in official documentation, include: injection site reactions, constipation, muscle cramps, vertigo, pruritus, and urticaria. Meanwhile other recipients of the therapy reported: nasopharyngitis, infection, sinusitis, fatigue, hypertension, nausea, arthralgia, back pain, and migraine. Due to potent vasodilative functions of CGRP, a list of contraindications was created. This list includes: manifestation of vascular diseases (myocardial infarction, unstable angina pectoris, stroke, transient ischemic attacks, coronary bypass surgery or other revascularization procedures within the last 12 months) and poorly controlled hypertension. It is still unknown what the potential course and prognosis of de novo myocardial infarction, cerebral ischemia and subarachnoid hemorrhage could be for patients receiving anti-CGRP medication. Calcitonin gene related peptide has been shown to promote angio- and lymphangiogenesis. Post-ischemic angiogenesis has been observed with the release of CGRP. Meanwhile, CGRP has been shown to improve lymphangiogenesis in secondary lymphedema. Further warnings concerning pregnancy and the desire to have children, potential damage to the blood-brain barrier (e.g. meningitis, stroke, after neurosurgery) and recent peripheral nerve lesions have arisen; and, appropriate longitudinal observations are only now being reported.

While autonomic symptoms of migraine are well known - such as: nausea/vomiting, hyperhidrosis, pallor, palpitations, and lightheadedness - the methods with which earlier investigations evaluated them are not as well-standardized. A review by Miglis, from 2018, summarizes that most studies of autonomic function in migraine showed reduced sympathetic function in migraineurs; while others, reported increased sympathetic function; and others still, showed normal sympathetic function. Likewise, the majority of studies reported normal parasympathetic cardiovagal function; while others, reported decreased parasympathetic function. Miglis goes on to describe in his review, a variety of investigations used to arrive at these conclusions - heart rate variability (HRV) studies, autonomic cardiovascular reflex testing and imagining studies. These paradoxical results can be interpreted as being caused by methodological inconsistency between investigations. For example, some HRV investigations elect to use 24h continuous electrocardiogram (ECG) monitoring, while others use ECG measurements during the head-up tilt test to gather HRV data. This results in the uncoordinated use of different methods, which ultimately illustrates the need for consistent, standardized testing of the ANS in migraine studies.

Considering the concerns expressed by Tringali and Navarra - to observe the long-term effects of CGRP-inhibition, as it pertains to autonomic function - there currently exists great potential to address this gap in knowledge. Therefore, this non-therapeutic biomedical study aims to address this lack of literature, by obtaining and comparing standardized healthy CAD values with those of migraineurs, observing CAD values in migraine patients off prophylactic therapy - in both the ictal and peri-ictal phases of the migraine cycle - and then comparing baseline CAD values with CAD values during anti-CGRP therapy.

Primary explorative questions:

This study will aim to address the autonomic aspects of migraine, through a newly published objective autonomic function scoring. It aims to explore whether differences exist in the autonomic function values (CAD) between healthy people and migraine patients. Furthermore, it will aim to explore the CAD differences between migraine attack-phases (peri-ictal and interictal). Lastly, over the course of 5 months, this study will explore whether inhibition of CGRP - as an anti-CGRP-mAb class-effect - affects these autonomic function scores. The following questions will be answered:

Q1: Is there a difference in CAD values between healthy controls and migraine patients off prophylactic medication?

Q2: Is there a difference in the CAD values of migraine patients during a migraine attack (peri-ictal phase) and their respective CAD values between attacks (interictal phase)?

Q3: Is there a difference in CAD values of migraine patients before anti-CGRP treatment and during treatment with anti-CGRP-mAbs (class effect on autonomic functions)?

Secondary Question:

To support the examination of these three questions, validated questionnaires will be used to assess the subjective effect of anti-CGRP-mAbs on: monthly migraine and headache days, autonomic function, quality of life and psychiatric symptoms.

Study Proceudres:

For the patients the study will comprise of: 1) a patient screening phase (following recruitment); 2) two clinical baseline visits (day 0 and one day between days 1 and 30); 3) an evaluation visit (month 5), which will also serve as the End of Study (EOS); and 4) a telephone follow-up. For the healthy controls the study will comprise: 1) a patient screening phase; 2) one testing visit (day 0); and 3) a telephone follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Chronic migraine according to ICHD-3
* Episodic migraine without aura or with aura according to ICHD-3
* Unsuccessful treatment with 3 or more established prophylactic drugs
* Medicine costs are covered by health insurance
* Healthy controls must be free from any diagnosed chronic disease or acute infection requiring medication

Exclusion Criteria:

* Pregnancy and lactation
* Neurosurgical interventions performed within the last 12 months
* Coronary bypass surgery or revascularization procedures performed within the last 12 months
* History of transient ischemic attacks (TIA), stroke, stable or unstable angina pectoris, myocardial infarction or uncontrolled hypertension
* Known hypersensitivity to therapy with an anti-CGRP Antibodies
* History of a disorder (other than migraine) that may affect the results of autonomic tests
* Healthy controls must have no personal or family history of migraine

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients diagnosed to be suffering from migraine without aura, migraine with aura or chronic migraine according to the diagnostic criteria of the International Classification of Headache Disorders, third edition (ICHD-3). Patients will be ages 18 to 64. It is mandatory they have valid health insurance provided by one of the insurance institutions of Austria.
  Controls must be healthy (free of any diagnosed chronic disease or acute infection requiring medication), chosen to be as similar as possible to migraine patients, in terms of age and sex
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from Day 0 Cardiovagal Autonomic Dysfunction (CAD) at 5 months | Day 0, Month 5 (EOS)
  It is derived from the Composite Autonomic severity scale (CASS), an "unbiased and full quantification" of the autonomic functions in the cardiovagal, adrenergic and sudomotor domain. The total CASS score has "a direct clinical meaning since it ranks the generalized dysautonomia as mild, moderate and severe". By isolating two of the indices of the CASS - adrenergic index (AI) and cardiovagal index (CI) - one can quantify the Cardiovascular Autonomic Dysfunction (CAD). Results are referred to as normal (CAD total score = 0) or abnormal. Abnormal values are considered 1-7, indicating presence of CAD.
Change from Days 1-31 Cardiovagal Autonomic Dysfunction (CAD) at 5 months | Days 1-31, Month 5 (EOS)
  It is derived from the Composite Autonomic severity scale (CASS), an "unbiased and full quantification" of the autonomic functions in the cardiovagal, adrenergic and sudomotor domain. The total CASS score has "a direct clinical meaning since it ranks the generalized dysautonomia as mild, moderate and severe". By isolating two of the indices of the CASS - adrenergic index (AI) and cardiovagal index (CI) - one can quantify the Cardiovascular Autonomic Dysfunction (CAD). Results are referred to as normal (CAD total score = 0) or abnormal. Abnormal values are considered 1-7, indicating presence of CAD.
Change from Days 0 Cardiovagal Autonomic Dysfunction (CAD) at Days 1-31 | Day 0, Days 1-31
  It is derived from the Composite Autonomic severity scale (CASS), an "unbiased and full quantification" of the autonomic functions in the cardiovagal, adrenergic and sudomotor domain. The total CASS score has "a direct clinical meaning since it ranks the generalized dysautonomia as mild, moderate and severe". By isolating two of the indices of the CASS - adrenergic index (AI) and cardiovagal index (CI) - one can quantify the Cardiovascular Autonomic Dysfunction (CAD). Results are referred to as normal (CAD total score = 0) or abnormal. Abnormal values are considered 1-7, indicating presence of CAD.

SECONDARY OUTCOMES:
Change from Days 0 Composite Autonomic Symptom Scale 31 (COMPASS-31) at 5 months | Day 0, Month 5 (EOS)
  The Composite Autonomic Symptom Scale 31 is a simplified autonomic symptom scoring scheme that follows a homogeneous pattern of scoring throughout the instrument. It quantifies 6 domains: Orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, bladder and pupillomotor functions. The 6 domains sum to a total COMPASS-31 score of 0 to 100. A higher score indicates greater autonomic impairment (worse score).
Change from Days 0 Day Impact Questionnaire (HIQ) at 5 months | Day 0, Month 5 (EOS)
  The Headache Impact Questionnaire is a six-item questionnaire which provides group-level comparisons, patient-level screening, and is responsive to changes in impact of days with headache. The HIQ items cover a substantial range of headache impact as defined by a much larger pool of items and include content areas found in most widely used tools for measuring headache impact. The 6 items sum to a total HIQ score of 0 to 24. A higher score indicates a greater burden of headache (worse score).
Change from Days 0 Non-Headache Day Impact Questionnaire (Non-HIQ) at 5 months | Day 0, Month 5 (EOS)
  The Non-Headache Day Impact Questionnaire is a six-item questionnaire which provides group-level comparisons, patient-level screening, and is responsive to changes in days without headache. The 6 items sum to a total non-HIQ score of 0 to 24. A higher score indicates a greater burden on headache-free days (worse score).
Change from Days 0 Migraine Disability Assessment Scale (MIDAS) at 5 months | Day 0, Month 5 (EOS)
  The Migraine Disability Assessment Scale is a 5-item self-administered questionnaire. It is used to quantify headache-related disability; and, has been shown as highly reliable in population-based samples of migraine headache sufferers. The score is the sum total of days affected by migraine. The 5 items sum to a total MIDAS score of 0 to 155. A higher score indicates greater headache-related disability (worse score).
Change from Days 0 Depression Anxiety Stress Scale (DASS) at 5 months | Day 0, Month 5 (EOS)
  The Depression Anxiety Stress Scale is a set of three self-report scales designed to measure the negative emotional states of depression, anxiety and stress. The DASS was constructed to further the process of defining, understanding, and measuring the pervasive and clinically significant emotional states usually described as depression, anxiety and stress. The 21-item sum is multiplied by a factor of 2, to result in a total DASS score of 0 to 126. Scoring is used to discriminate between the three related states of depression, anxiety and stress; with a higher score indicating greater indication of the three emotional states (worse score).

CONTACTS AND LOCATIONS:
Overall Officials: Christian Wöber, Prof. MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GBD 2017 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 354 diseases and injuries for 195 countries and territories, 1990-2017: a systematic analysis for the Global Burden of Disease Study 2017. Lancet. 2018 Nov 10;392(10159):1789-1858. doi: 10.1016/S0140-6736(18)32279-7. Epub 2018 Nov 8. PMID 30496104
- [Background] Miglis MG. Migraine and Autonomic Dysfunction: Which Is the Horse and Which Is the Jockey? Curr Pain Headache Rep. 2018 Feb 23;22(3):19. doi: 10.1007/s11916-018-0671-y. PMID 29476276
- [Background] Headache Classification Committee of the International Headache Society (IHS) The International Classification of Headache Disorders, 3rd edition. Cephalalgia. 2018 Jan;38(1):1-211. doi: 10.1177/0333102417738202. No abstract available. PMID 29368949
- [Background] Sacks O. Migraine: The evolution of a common disorder. 1st ed. Univ of California Press, 1970, p. 53-205.
- [Background] Cernuda-Morollon E, Martinez-Camblor P, Alvarez R, Larrosa D, Ramon C, Pascual J. Increased VIP levels in peripheral blood outside migraine attacks as a potential biomarker of cranial parasympathetic activation in chronic migraine. Cephalalgia. 2015 Apr;35(4):310-6. doi: 10.1177/0333102414535111. Epub 2014 May 20. PMID 24847167
- [Background] Mosek A, Novak V, Opfer-Gehrking TL, Swanson JW, Low PA. Autonomic dysfunction in migraineurs. Headache. 1999 Feb;39(2):108-17. doi: 10.1046/j.1526-4610.1999.3902108.x. PMID 15613203
- [Background] Russell FA, King R, Smillie SJ, Kodji X, Brain SD. Calcitonin gene-related peptide: physiology and pathophysiology. Physiol Rev. 2014 Oct;94(4):1099-142. doi: 10.1152/physrev.00034.2013. PMID 25287861
- [Background] Low PA. Testing the autonomic nervous system. Semin Neurol. 2003 Dec;23(4):407-21. doi: 10.1055/s-2004-817725. PMID 15088262
- [Background] Buijs RM, Swaab DF, editors. Testing the autonomic nervous system. In: Handbook of clinical neurology Autonomic nervous system. vol. 117. Elsevier, 2013, pp.115-136.
- [Background] Novak P. Quantitative autonomic testing. J Vis Exp. 2011 Jul 19;(53):2502. doi: 10.3791/2502. PMID 21788940
- [Background] Hansen JM, Schankin CJ. Cerebral hemodynamics in the different phases of migraine and cluster headache. J Cereb Blood Flow Metab. 2019 Apr;39(4):595-609. doi: 10.1177/0271678X17729783. Epub 2017 Aug 31. PMID 28857642
- [Background] Chong CD, Schwedt TJ, Hougaard A. Brain functional connectivity in headache disorders: A narrative review of MRI investigations. J Cereb Blood Flow Metab. 2019 Apr;39(4):650-669. doi: 10.1177/0271678X17740794. Epub 2017 Nov 20. PMID 29154684
- [Background] Messina R, Filippi M, Goadsby PJ. Recent advances in headache neuroimaging. Curr Opin Neurol. 2018 Aug;31(4):379-385. doi: 10.1097/WCO.0000000000000573. PMID 29952833
- [Background] Tringali G, Navarra P. Anti-CGRP and anti-CGRP receptor monoclonal antibodies as antimigraine agents. Potential differences in safety profile postulated on a pathophysiological basis. Peptides. 2019 Jun;116:16-21. doi: 10.1016/j.peptides.2019.04.012. Epub 2019 Apr 21. PMID 31018157
- [Background] Deen M, Correnti E, Kamm K, Kelderman T, Papetti L, Rubio-Beltran E, Vigneri S, Edvinsson L, Maassen Van Den Brink A; European Headache Federation School of Advanced Studies (EHF-SAS). Blocking CGRP in migraine patients - a review of pros and cons. J Headache Pain. 2017 Sep 25;18(1):96. doi: 10.1186/s10194-017-0807-1. PMID 28948500
- [Background] Ko JA, Mizuno Y, Ohki C, Chikama T, Sonoda KH, Kiuchi Y. Neuropeptides released from trigeminal neurons promote the stratification of human corneal epithelial cells. Invest Ophthalmol Vis Sci. 2014 Jan 7;55(1):125-33. doi: 10.1167/iovs.13-12642. PMID 24327615
- [Background] He H, Chai J, Zhang S, Ding L, Yan P, Du W, Yang Z. CGRP may regulate bone metabolism through stimulating osteoblast differentiation and inhibiting osteoclast formation. Mol Med Rep. 2016 May;13(5):3977-84. doi: 10.3892/mmr.2016.5023. Epub 2016 Mar 21. PMID 27035229
- [Background] Mizutani T, Yokoyama Y, Kokuryo T, Kawai K, Miyake T, Nagino M. Calcitonin gene-related peptide regulates the early phase of liver regeneration. J Surg Res. 2013 Jul;183(1):138-45. doi: 10.1016/j.jss.2012.11.028. Epub 2012 Dec 1. PMID 23218524
- [Background] Holzmann B. Antiinflammatory activities of CGRP modulating innate immune responses in health and disease. Curr Protein Pept Sci. 2013 Jun;14(4):268-74. doi: 10.2174/13892037113149990046. PMID 23745695
- [Background] Kee Z, Kodji X, Brain SD. The Role of Calcitonin Gene Related Peptide (CGRP) in Neurogenic Vasodilation and Its Cardioprotective Effects. Front Physiol. 2018 Sep 19;9:1249. doi: 10.3389/fphys.2018.01249. eCollection 2018. PMID 30283343
- [Background] Robertson CE. Could CGRP Antagonists Be Helpful in the Fight Against COVID-19? Headache. 2020 Jul;60(7):1450-1452. doi: 10.1111/head.13853. Epub 2020 Jun 15. No abstract available. PMID 32386433
- [Background] Tepper SJ. Anti-Calcitonin Gene-Related Peptide (CGRP) Therapies: Update on a Previous Review After the American Headache Society 60th Scientific Meeting, San Francisco, June 2018. Headache. 2018 Nov;58 Suppl 3:276-290. doi: 10.1111/head.13417. PMID 30403405
- [Background] Szperka CL, VanderPluym J, Orr SL, Oakley CB, Qubty W, Patniyot I, Lagman-Bartolome AM, Morris C, Gautreaux J, Victorio MC, Hagler S, Narula S, Candee MS, Cleves-Bayon C, Rao R, Fryer RH, Bicknese AR, Yonker M, Hershey AD, Powers SW, Goadsby PJ, Gelfand AA. Recommendations on the Use of Anti-CGRP Monoclonal Antibodies in Children and Adolescents. Headache. 2018 Nov;58(10):1658-1669. doi: 10.1111/head.13414. Epub 2018 Oct 15. No abstract available. PMID 30324723
- [Background] Robbins L. CGRP Antagonists: Physiologic Effects and Serious Side Effects. Headache. 2018 Oct;58(9):1469-1471. doi: 10.1111/head.13408. Epub 2018 Oct 11. No abstract available. PMID 30308092
- [Background] Feuerstein M, Bush C, Corbisiero R. Stress and chronic headache: a psychophysiological analysis of mechanisms. J Psychosom Res. 1982;26(2):167-82. doi: 10.1016/0022-3999(82)90034-4. PMID 7077548
- [Background] Ewing DJ, Martyn CN, Young RJ, Clarke BF. The value of cardiovascular autonomic function tests: 10 years experience in diabetes. Diabetes Care. 1985 Sep-Oct;8(5):491-8. doi: 10.2337/diacare.8.5.491. PMID 4053936
- [Background] Treister R, O'Neil K, Downs HM, Oaklander AL. Validation of the composite autonomic symptom scale 31 (COMPASS-31) in patients with and without small fiber polyneuropathy. Eur J Neurol. 2015 Jul;22(7):1124-30. doi: 10.1111/ene.12717. Epub 2015 Apr 23. PMID 25907824
- [Background] Matei D, Constantinescu V, Corciova C, Ignat B, Matei R, Popescu CD. Autonomic impairment in patients with migraine. Eur Rev Med Pharmacol Sci. 2015 Oct;19(20):3922-7. PMID 26531280
- [Background] Piovesan EJ, Sobreira CF, Scola RH, Lorenzoni PJ, Lange MC, Werneck LC, Smith D, Silberstein S. Episodic migraine associated with postural orthostatic tachycardia syndrome and vasovagal syncope: migraine triggers neuromediated syncope. Arq Neuropsiquiatr. 2008 Mar;66(1):77-9. doi: 10.1590/s0004-282x2008000100018. No abstract available. PMID 18392420
- [Background] Rauschel V, Straube A, Suss F, Ruscheweyh R. Responsiveness of the autonomic nervous system during paced breathing and mental stress in migraine patients. J Headache Pain. 2015;16:82. doi: 10.1186/s10194-015-0567-8. Epub 2015 Sep 16. PMID 26377932
- [Background] Cambron M, Maertens H, Paemeleire K, Crevits L. Autonomic function in migraine patients: ictal and interictal pupillometry. Headache. 2014 Apr;54(4):655-62. doi: 10.1111/head.12139. Epub 2013 Jun 28. PMID 23808550
- [Background] Rossato A, Veronese F, Maggioni F, Vedovetto V, Zancan A, Biasiolo M, Bilora F. Autonomic dysfunction and endothelial changes in migraine sufferers. Panminerva Med. 2011 Mar;53(1):13-8. PMID 21346700
- [Background] Pogacnik T, Sega S, Pecnik B, Kiauta T. Autonomic function testing in patients with migraine. Headache. 1993 Nov-Dec;33(10):545-50. doi: 10.1111/j.1526-4610.1993.hed3310545.x. PMID 8294192
- [Background] Benjelloun H, Birouk N, Slaoui I, Coghlan L, Bencheikh BO, Jroundi I, Benomar M. [Autonomic profile of patients with migraine]. Neurophysiol Clin. 2005 Oct;35(4):127-34. doi: 10.1016/j.neucli.2005.06.001. Epub 2005 Sep 29. French. PMID 16311208
- [Background] Crnosija L, Krbot Skoric M, Andabaka M, Junakovic A, Martinovic V, Ivanovic J, Mesaros S, Pekmezovic T, Drulovic J, Habek M. Autonomic dysfunction in people with neuromyelitis optica spectrum disorders. Mult Scler. 2020 May;26(6):688-695. doi: 10.1177/1352458519837703. Epub 2019 Mar 19. PMID 30887872
- [Background] Sletten DM, Suarez GA, Low PA, Mandrekar J, Singer W. COMPASS 31: a refined and abbreviated Composite Autonomic Symptom Score. Mayo Clin Proc. 2012 Dec;87(12):1196-201. doi: 10.1016/j.mayocp.2012.10.013. PMID 23218087
- [Background] Kosinski M, Bayliss MS, Bjorner JB, Ware JE Jr, Garber WH, Batenhorst A, Cady R, Dahlof CG, Dowson A, Tepper S. A six-item short-form survey for measuring headache impact: the HIT-6. Qual Life Res. 2003 Dec;12(8):963-74. doi: 10.1023/a:1026119331193. PMID 14651415
- [Background] Stewart WF, Lipton RB, Kolodner K, Liberman J, Sawyer J. Reliability of the migraine disability assessment score in a population-based sample of headache sufferers. Cephalalgia. 1999 Mar;19(2):107-14; discussion 74. doi: 10.1046/j.1468-2982.1999.019002107.x. PMID 10214536
- [Background] Lovibond, S.H. & Lovibond, P.F. (1995). Manual for the Depression Anxiety Stress Scales. (2nd. Ed.) Sydney: Psychology Foundation. ISBN 7334-1423-0.
- [Background] Peng KP, May A. Redefining migraine phases - a suggestion based on clinical, physiological, and functional imaging evidence. Cephalalgia. 2020 Jul;40(8):866-870. doi: 10.1177/0333102419898868. Epub 2020 Jan 13. PMID 31928343
- [Background] Schulte LH, May A. The migraine generator revisited: continuous scanning of the migraine cycle over 30 days and three spontaneous attacks. Brain. 2016 Jul;139(Pt 7):1987-93. doi: 10.1093/brain/aww097. Epub 2016 May 5. PMID 27190019
- [Background] Crnosija L, Krbot Skoric M, Lovric M, Junakovic A, Miletic V, Alfirev RS, Pavelic A, Adamec I, Habek M. Differences in neurohumoral and hemodynamic response to prolonged head-up tilt between patients with high and normal standing norepinephrine forms of postural orthostatic tachycardia syndrome. Auton Neurosci. 2017 Jul;205:110-114. doi: 10.1016/j.autneu.2017.05.007. Epub 2017 May 11. PMID 28522107
- [Background] Crnosija L, Krbot Skoric M, Adamec I, Lovric M, Junakovic A, Mismas A, Miletic V, Sprljan Alfirev R, Pavelic A, Habek M. Hemodynamic profile and heart rate variability in hyperadrenergic versus non-hyperadrenergic postural orthostatic tachycardia syndrome. Clin Neurophysiol. 2016 Feb;127(2):1639-1644. doi: 10.1016/j.clinph.2015.08.015. Epub 2015 Sep 4. PMID 26386646
- [Background] Heart rate variability: standards of measurement, physiological interpretation and clinical use. Task Force of the European Society of Cardiology and the North American Society of Pacing and Electrophysiology. Circulation. 1996 Mar 1;93(5):1043-65. No abstract available. PMID 8598068
- [Background] Yoshida S, Tanaka H, Mizutani M, Nakao R, Okamoto N, Kajiura M, Kanbara Y, Tamai H. Autonomic nervous system function in adolescent migraineurs. Pediatr Int. 2017 Sep;59(9):991-995. doi: 10.1111/ped.13342. PMID 28612516
- [Background] Bates D et al. Fitting Linear Mixed-Effects Models Using lme4. Journal of Statistical Software 2015; 67, 1: 1-48. https://doi.org/10.18637/jss.v067.i01.
- [Background] R Core Team. R: A language and environment for statistical computing. R Foundation for Statistical Computing, Vienna, Austria. (2014). URL http://www.R-project.org/
- [Background] SAS Institute Inc. Base SAS® 9.4 Procedures Guide. Cary, NC: SAS Institute Inc. (2011). URL: http://documentation.sas.com/?docsetId=acadbas&docsetTarget =acadbas.pdf&docsetVersion=9.4&locale=en